CLINICAL TRIAL: NCT05788003
Title: Female Genital Schistosomiasis in Tanzania: Evaluation of Prevalence and Performance of Schistosoma Haematobium-specific Polymerase Chain Reaction (PCR) on Operator-based and Self-collected Cervical-vaginal Samples Among Women Living in Endemic Areas, North-western Tanzania
Brief Title: Female Genital Schistosomiasis in Tanzania
Acronym: ShWAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-07
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Schistosomiasis Mansoni
Keywords: Female Genital Schistosomiasis
MeSH Terms: conditions — Schistosomiasis mansoni

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: self-collected and operator-collected swab followed by molecular analysis — A single midday urine sample and two cervical-vaginal swabs (both self-collected and speculum-aided collected by a female healthcare worker) will be obtained from participating women and processed using urine filtration and polymerase chain reaction (PCR) for cervico-vaginal samples.

SUMMARY:
A cross-sectional survey will be conducted among 200 volunteering women aged 18- 45 years and having had prior sexual activity living in the target villages of Itilima and Maswa districts, North-western Tanzania. A single midday urine sample and two cervical-vaginal swabs (both self-collected and speculum-aided collected by a female healthcare worker) will be obtained from participating women and processed using urine filtration and polymerase chain reaction (PCR) for cervico-vaginal samples. A pre-tested structure questionnaire will be used to collect sociodemographic, clinical, and sampling acceptability information from participants.

DETAILED DESCRIPTION:
A cross-sectional survey will be conducted among 200 volunteering women aged 18-45 years and having had prior sexual activity living in the target villages of Itilima and Maswa districts, North-western Tanzania. A single midday urine sample and two cervical-vaginal swabs (both self-collected and speculum-aided collected by a female healthcare worker) will be obtained from participating women and processed using urine filtration and polymerase chain reaction (PCR) for cervico-vaginal samples. A pre-tested structure questionnaire will be used to collect sociodemographic, clinical, and sampling acceptability information from participants. Prevalence of Female Genital Schistosomiasis (FGS) will be estimated based on positivity of at least one genital specimen. Quantitative data will be described using means/medians and standard deviation/interquartile range, as appropriate. Qualitative data will be described as numbers and percentages, and compared using Chi-squared or Fisher Exact test, as appropriate. Sensitivity of the two genital sampling methods will be compared using the composite reference constituted by positivity in at least one genital swab, and the performance of the two methods compared using Cohen's Kappa statistics, Fisher's Exact test and parametric/nonparametric test for comparison of PCR Ct values, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years,
* having had prior sexual activity (to allow speculum-aided gynaecological visit and genital sampling),
* resident in any of the selected village of Itilima and Maswa districts,
* irrespective of complaining of urogenital symptoms,
* not reporting any exclusion criteria,
* willing to participate to the study as documented by signing the informed consent form.

Exclusion Criteria:

* Menstruation at the time of visit (since this limits visualization of the cervix and correct sampling);
* no prior sexual activity (since this does not allow the use of a speculum in the visit);
* known pregnancy;
* documented treatment for schistosomiasis in the past 6 months;
* age <18 or >45 years;
* unwilling to sign the informed consent form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-03-17 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Female Genital Schistosomiasis | 6 months
  Prevalence of Female Genital Schistosomiasis among women aged 18-45 years living in selected villages of Itilima and Maswa districts, North-western Tanzania

SECONDARY OUTCOMES:
Acceptability of different sample collection and diagnostic approaches (genital self-sampling, speculum-aided collected genital sampling conducted by female or hypothetically by male healthcare workers) | 6 months
  The participant will be asked some questions about her clinical history and about her experience with self-sampling.
Sensitivity and specificity of self-collected versus healthcare operator speculum-aided collected cervico-vaginal samples for diagnosis of Female Genital Schistosomiasis | 6 months
  Sensitivity of the two genital sampling methods will be calculated using the composite reference constituted by positivity in at least one genital swab, and the performance of the two methods.

CONTACTS AND LOCATIONS:
Locations (2):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy
- Catholic University of Health and Allied Sciences (CUHAS), Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared together with the paper describing the study results.